CLINICAL TRIAL: NCT06441669
Title: Effect of Letermovir Prophylaxis on Cytomegalovirus-specific Immune Reconstitution Post Unrelated Cord Blood Transplantation
Brief Title: Effect of Letermovir Prophylaxis on CMV-specific Immune Reconstitution Post UCBT
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: CBCMV001
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Cytomegalovirus Infection Reactivation
Keywords: Cytomegalovirus Infection; Umbilical Cord Blood Transplantation; CMV-Specific Immune Reconstitution; Letermovir
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- letermovir group: Patients will be given Letermovir with a recommended dose of 480 mg per day (or 240 mg per day in patients taking cyclosporine or according to clinical instructions) from +1 day to +100 days after UCBT.
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Patients will be given Letermovir with a recommended dose from +1 day to +100 days after UCBT.

SUMMARY:
To explore the effect of letermovir prophylaxis on cytomegalovirus-specific immune reconstitution post unrelated cord blood transplantation

DETAILED DESCRIPTION:
To explore the effect of letermovir prophylaxis on cytomegalovirus-specific and other lymphocyte subsets immune reconstitution post unrelated cord blood transplantation, and to analyze the potential mechanism and risk factors of late CMV reactivation after letermovir discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Patients are receiving a first unrelated cord blood transplantation (UCBT).
* Patients start letemovir prophylaxis within 0-28 days post UCBT.

Exclusion Criteria:

* Patients having active CMV DNAemia at the time of letermovir initiation.
* Patients recruited in a clinical study on an anti-CMV trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study consists 60 cases recipients of UCBT. All patients will receive letermovir prophylaxis within 0-28 days post UCBT.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Numbers of immune cells in peripheral blood | one year
  PBMCs from UCBT recipients were collected at 1 month, 2 month, 3 month, and 6 month and 12 month after HSCT, and tested for CMV-specific T cells, NK cells, T cells and other subsets.
CMV DNAemia | one year
  CMV DNAemia is defined as the detection of CMV DNA in samples of plasma, whole blood or isolated peripheral blood leukocyte.
Incidence of refractory CMV infection | one year
  Refractory CMV infection is defined as CMV viral load remaining at the same level or increasing despite appropriately doses of antiviral therapy for at least 2 weeks
late CMV reactivation | one year
  Late CMV reactivation is defined as reactivation that occurs 100 days post UCBT, which means reactivation after discontinuing LET prophylaxis.

SECONDARY OUTCOMES:
Treatment-ralated mortality | one year
  Treatment-ralated mortality
Incidence of other viral infection and viral-associated disease | one year
  Other viral infection and viral-associated diseases including EBV, ADV, HHV-6, BKV and HSV
Overall survival | one year
  Overall survival
serum immunoglobulin assay | 1,3,6,9 month post UCBT
  The serum levels of IgG, IgM, and IgA were measured

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, ph.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China (Anhui Provicial Hospital)
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China